CLINICAL TRIAL: NCT04445233
Title: The COVID-19 Household Transmission Study (CO-HOST) - Epidemiology of SARS-CoV-2 Transmission Within the Household
Brief Title: COVID-19 Household Transmission Study
Acronym: CO-HOST
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 20-0982; 550KR242023 (Other Grant/Funding Number: NIH)
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: COVID-19
Keywords: Household; COVID-19; Coronavirus; Infection; Transmission; SARS-CoV-2; Nasopharyngeal; Nasal Swabs
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — nasopharyngeal swabs, nasal swabs, nasal strips, blood samples, saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- COV Participants: COVID-positive index cases (COV): Participants who are greater than or equal to 18 years of age who test positive for COVID-19 by positive NP swab
  Interventions: Device: COVID-19 IgM-IgG Rapid Test
- COV-HC Participants: Household contact of COVID-positive index case (COV-HC): Household contacts greater than 1 year of age currently living in the same home as the COVID-positive index case
  Interventions: Device: COVID-19 IgM-IgG Rapid Test

INTERVENTIONS:
Device: COVID-19 IgM-IgG Rapid Test — Used to detect the IgG and IgM antibodies of the novel coronavirus in human whole blood (capillary or venous), serum, or plasma.

SUMMARY:
This study will test and follow persons quarantined at home after testing positive for SARS-CoV-2 (COV) aged 18 years and older and their household members aged 1 year and older.

The purpose of this research study is to understand how often COVID-19 (Coronavirus Disease 2019) spreads in the household when someone who tests positive for the virus self-isolates at home.

The purpose of the extension part of the study is to help us understand long-term immunity to COVID-19. We are interested in how our immune system might still protect us from COVID-19 even after antibody levels decrease or are no longer detected. We are also interested in how immunity to COVID-19 is different in kids vs. adults.

DETAILED DESCRIPTION:
This study will enroll approximately 200 men and women ≥ 18 years of age who are SARS-CoV-2 PCR positive undergoing home quarantine & approximately 200-1500 immediate household contacts, both male and female, ≥ 1 year of age.

This study will test and follow persons quarantined at home after testing positive for SARS-CoV-2 (COV) and their household members.

The CO-HOST mobile nurse initiates a home visit to the home of the COVID-19 index case after they and their household members (COV-HC) verbally express interest in the study and provide consent or assent as appropriate. At the first visit, nasopharyngeal (NP) swabs and blood are collected from COV and all members of the household (COV-HC) to determine infection status. Additional samples (nasal swabs, saliva, nasal strips), both nurse-collected and self-collected, may also be collected from COV and COV-HC. The nurse will provide specific instructions and training on how to perform self-collected swabs.

Every week, thereafter, COV-HC are tested during the 28 days of the study. If home visits are not possible, then participants will perform self-collected swabs for testing. If COV-HC develops symptoms, they will be referred per standard of care (SOC).

If COV or COV-HC are hospitalized, they will remain in the study for outcome assessment, but without further sample collections.

As part of the extension to the study, the study team will come back to previous enrolled participants' houses for a single visit at about 6 months from when they enrolled in this study. If these participants prefer, they could come to UNC for this visit instead. At this visit, the study team will collect these participants' blood sample and draw up to 10 tsp of blood. The study team will also perform a COVID-19 rapid antibody test, which uses two-three drops of blood from a finger prick. These participants will also be asked to complete a short (5-minute) online questionnaire.

After this visit, if these participants have not already been vaccinated, then the study team will give them the option to participate in one more visit at their house or at UNC within 1-3 months after they receive the COVID vaccine to collect a blood sample (up to 10 tsp). The study team will also repeat the rapid antibody test with another finger prick.

ELIGIBILITY:
Inclusion Criteria:

COVID-positive index cases (COV):

* Any patient greater than or equal to18 years of age with a positive qualitative nasopharyngeal or nasal swab for SARS-CoV-2 obtained at UNC Hospitals or an outpatient clinic
* COVID-19 diagnosis by positive NP swab
* Willingness to self-isolate at home for a 14-day period
* Living with at least one household contact who is also willing to consent to study follow-up
* Living within reasonable driving distance (<1 hour) suitable for home visits by study team

Household contact of COVID-positive index case (COV-HC):

• Household contacts greater than 1 year of age currently living in the same home as the COVID-positive index case without plans to leave to live elsewhere through the end of the 28-day study.

Exclusion Criteria:

COVID-positive index cases (COV): None

Household contact of COVID-positive index case (COV-HC):

• Previously participated in this study (as index case or household contact)

For the extension part of CO-HOST, study participants greater than 65 years of age who tested positive for acute SAR-CoV-2 infection by PCR or seroconversion (antibody status became positive) during their participation in the first month of the study, will be eligible. They will be excluded if they previously received immunologic therapy (i.e., exogenous anti-SARS-CoV-2 monoclonal antibodies) for COVID-19 infection.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Men and women ≥ 18 years of age who are SARS-CoV-2 PCR positive undergoing home quarantine & immediate household contacts, both male and female, ≥ 1 year of age will all be asked to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Number of Households with New SARS-CoV-2 Infection by Day 28 | 28 days
  Secondary household infection rate
Risk Factors Associated with Secondary Household Transmission | 28 days
  Secondary household infection rate risk factors

SECONDARY OUTCOMES:
Number of Self-Swab Tests vs. NP Swabs at Day 1 with Detectable Viral Load | 1 day
  Sensitivity of self-collected nasal swabs

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Lin, MD, MSCR, Principal Investigator — UNC-Chapel Hill
Locations (1):
- University of North Carolina Health Care, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data that supports the results will be shared beginning 12 to 24 months following publication provided the investigator/researcher who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: 12-24 months after publication
Access Criteria: Investigators/researchers who propose to use study data will need to have IRB, IEC, or REB approval and an executed data use/sharing agreement with UNC.